CLINICAL TRIAL: NCT07068789
Title: Revascularization of Single Versus Multiple Infrapopliteal Vesseles in Chronic Limb Threatening Ischemia : Limb Salvage Rate
Brief Title: Revascularization of Single Vesrus Multiple Infrapopliteal Vessels in Chronic Limb Threatening Ischemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelrahman Hafez, Mahmoud Abdelrahman Hafez, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-6-14MS
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Chronic Limb Threatening Ischemia; Infrapopliteal Arterial Occlusive Disease
Keywords: chronic limb threatening ischemia; infrapopliteal arteries angioplasty; limb salvage; endovascular revascularization
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty, Balloon

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel groups based on the revascularization strategy received : single vessel infrapopliteal angioplasty or multiple vessel infrapoplital angioplasty . Each participant will remain in the same intervention group throughout the study period and outcomes will be comapred between the two groups
Masking Description: due to nature of the intervention procedures masking was not feasible the number of infrapopliteal arteries treated is clearly documented in procedural reports and imaging and therefore both participants and treating physicians were aware of the assigned intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- three vessel revascularization (Experimental): patients in this group will undergo will receive angioplasty of all three infrapopliteal arteries
  Interventions: Procedure: balloon angioplasty
- two vessel revascularization (Experimental): patients in this group will undergo will receive angioplasty of two infrapopliteal arteries
  Interventions: Procedure: balloon angioplasty
- single vessel revascularization (Experimental): patients in this group will undergo will receive angioplasty of only one infrapopliteal artery
  Interventions: Procedure: balloon angioplasty

INTERVENTIONS:
Procedure: balloon angioplasty — endovascular angioplasty of infrapopliteal arteries performed using standard balloon catheters under fluroscopic guidance to restore blood flow to the ischemic area

SUMMARY:
This interventional prospective study aims to assess the effectiveness of single vessel versus multiple vessel infrapopliteal angioplasty in patients with chronic threatening limb ischemia . The study compares limb salvage rates and clinical outcomes across two groups over a defined follow up period

ELIGIBILITY:
Inclusion Criteria: 1. patients aged 40 years or older 2. patients with Rutherford category "4" and "5" 3. patients with angiographic evidence of infrapopliteal vessel occlusive disease -

Exclusion Criteria:

1. patients who refuse to participate in the study
2. patients with isolated proximal arterial disease (e.g SFA or popliteal ) without infrapopliteal involvement
3. patients who develop acute thrombosis , flow limiting dissection or perforation in the infrapopliteal arteries during intervention -

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
limb salvage rate | 6 months ( with optional follow up at 12 months )
  percentage of patients who remain free from major lower limb amputation during the period of follow up after angioplasty
limb salvage rate | 6 months ( with optional follow up at 12 months )
  percentage of patients who avoid major amputation during the period of follow up following angioplasty procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of Sohag, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
not applicable data will be used internally for academic purpose only